CLINICAL TRIAL: NCT01252784
Title: Reduced-intensity Conditioning Allogeneic Hematopoietic Cell Transplantation Followed by Prophylactic Dose-escalating Donor Lymphocyte Infusions in Higher Risk Myelodysplastic Syndrome
Brief Title: Reduced-intensity Conditioning Allogeneic Hematopoietic Cell Transplantation
Acronym: RICandDLI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Other Study IDs: Allo-039
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: higher risk MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — This clinical trial will use busulfan, fludarabine, thymoglobulin and methylprednisolone for conditioning therapy, and cyclosporine and methotrexate for prevention of GVHD. All drugs had been previously accepted for administration to human in respective indication and there is no need to further evaluate the efficacy and the safety of each drug separately. Dose-escalating DLI is also widely accepted procedure after allogeneic HCT.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the feasibility and efficacy of reduced-intensity conditioning allogeneic HCT followed by prophylactic dose-escalating DLIs in patients with higher risk MDS.

DETAILED DESCRIPTION:
Conditioning therapy

* Busulfan 3.2 mg/kg/d on d-7 to -6
* Fludarabine 30 mg/m2 on d-7 to -2
* ATG 1.5-3.0 mg/kg/d on d-3 to -1
* Methylpred 2 mg/kg/d on d-4 to -1

Mobilization and harvest

* Donor
* G-CSF 10 mcg/kg/d s.c. on d-3 to 0
* Harvest of PBMCs on d 0 to +1

Infuse G-PBMCs on d 0 to d+1.

* Donor G-PBMC infusion

GVHD prophylaxis

* Cyclosporine 1.5 mg/kg i.v. q 12 hrs beginning on d-1 and changed to oral dosing (with twice the i.v. dose) when oral intake is possible. Tapered beginning between d+30 and d+60.
* Methotrexate 15 mg/m2 i.v. on d+2, and 10 mg/m2 i.v. on d+4 and d+7

Prophylactic dose-escalating DLIs

* Begin at d+120 or at least 2 wks after IST discontinuation.
* No evidence of recurrence or GVHD CD3+ cell dose increment q 4 wks 4Three dose levels

ELIGIBILITY:
Inclusion Criteria:

1. Patients with higher risk MDS including chronic myelomonocytic leukemia

   * RAEB-1 or RAEB-2
   * IPSS Intermediate-2 or High risk category
   * Chronic myelomonocytic leukemia
2. Patients with appropriate hematopoietic cell donor

   * HLA-matched sibling
   * HLA-matched unrelated donor
   * HLA-mismatched familial donor 3.16 years old or older

Exclusion Criteria:

* • Presence of significant active infection

  * Presence of uncontrolled bleeding
  * Any coexisting major illness or organ failure
  * Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with higher risk MDS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
relapse incidence,duration of remission | 4years
  The efficacy of the treatment will be measured in terms of relapse incidence and duration of remission (the primary endpoints). The hematopoietic cell donors in the study will include HLA-matched sibling, HLA-matched unrelated donors, and HLA-mismatched familial donors.

SECONDARY OUTCOMES:
engraftment, donor chimerism, secondary graft failure,GVHD | 4 years
  •This study will evaluate engraftment, donor chimerism, secondary graft failure, acute and chronic graft-versus-host disease (GVHD), immune recovery, infections, non-relapse mortality, progression-free survival (PFS), and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- See also: Reduced-intensity conditioning allogeneic hematopoietic cell transplantation followed by prophylactic dose-escalating donor lymphocyte infusions in higher risk myelodysplastic syndrome — http://www.google.com